CLINICAL TRIAL: NCT01930903
Title: Proposing an Alternative Treatment to patiEnts for Whom DES Implantation is Not Indicated, Thanks to Pantera LUX Drug Eluting Balloon
Brief Title: PaneLux PTCA : Proposing an Alternative Treatment to patiEnts for Whom DES Implantation is Not Indicated, Thanks to Pantera LUX Drug Eluting Balloon
Acronym: PaneLux PTCA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Biotronik France (Industry)
Collaborators: MedPass International (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Purpose: Treatment
Other Study IDs: 201202
Record Dates: First submitted 2013-08-26; First posted 2013-08-29 (Estimated); Last update posted 2015-04-30 (Estimated); Status verified 2014-02

CONDITIONS: Coronary Artery Disease; High Bleeding Risk Patients
Keywords: PRO-Kinetic Energy BMS + Pantera Lux DEB combination
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Pantera Lux Drug Eluting Balloon — All patients are treated with the PRO-Kinetic Energy Stent and Pantera Lux drug eluting balloon for the last post dilatation.

SUMMARY:
The propose of this study is to demonstrate, whenever using Drug Eluting Stent is not possible, the clinical security at 12 months, of the combinaison Bare Metal Stent plus Drug Eluting Balloon.

ELIGIBILITY:
Inclusion Criteria:

1. Subject has provided a written informed consent
2. Subject >/= 18 years.
3. Patient affiliated to social security
4. Patient acceptable candidate who accept to be contacted at different terms of clinical follow up (1, 6 and 12 months)
5. Subject eligible for percutaneous coronary intervention AND undergoing a chronical oral anticoagulant treatment OR undergoing any semi-urgent invasive or non cardiac surgical planned intervention with major bleeding risks
6. Subject eligible for Dual Anti Platelet Therapy (DAPT) of acetyl salicylic acid and clopidogrel for at least 3 weeks
7. De Novo coronary lesions: >/= 50% - <100%
8. Subject, vessels and target lesion eligible for angioplasty with PRO-Kinetic Energy stent implantation and final post-dilatation with Pantera Lux drug eluting balloon.
9. Target lesion length </= 26 mm , visual estimation or by Quantitative Coronary Angiography (QCA)
10. Reference diameters targeted vessels >/=2.5mm and </= 4.0 mm (visual estimation or QCA)

Exclusion Criteria:

1. Pregnant or breast feeding females or females who intend to become pregnant during the time of the study
2. Subject with a life expectancy less than 1 year
3. Vulnerable subject, protected by law, unable to give his/her consent
4. Subject currently enrolled in other medical or drug study and has not reached the primary outcome measures of that study
5. Subject unable to be contacted for the clinical follow up at 1, 6 and 12 months
6. Subject under chronical oral anti-coagulant treatment (optionnal indication)
7. Subject undergoing any urgent invasive or surgical intervention with major bleeding risk, which can not maintain dual anti-platelet therapy (DAPT) for at least 3 weeks
8. In stent restenotic lesion
9. Target lesion on vessels with nominal diameter < 2.5 mm
10. Target lesion is located in or supplied by an arterial or venous bypass graft
11. Chronical Total occlusion (CTO)
12. Angioplasty indication for STEMI
13. Patient with signs of cardiogenic shock
14. Angioplasty antecedent with stent implantation (before 12 months for DES, before 6 months for BMS)
15. "Staged procedure" > 8 days after the initial angioplasty
16. Documented left ventricular ejection fraction (LVEF) </= 30%
17. Target lesion requiring before stent implantation a device other than a pre-dilatation balloon (including, but not only restricted to laser, cutting balloon, directional coronary atherectomy, rotational atherectomy etc…)
18. Known allergies to acetylsalicylic acid, active agent such Paclitaxel, Expicients like BHTC (Butiriltri-n-hexyl citrate), CoCr, Silicon Carbide.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2013-09; Primary Completion 2015-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Target Lesion Failure (TLF) at 12 months. | 12 months
  TLF is defined as a composite of cardiac death, any target vessel myocardial infarction (MI), urgent coronary artery bypass graft (CABG) and clinically driven target lesion revascularization (TLR).

SECONDARY OUTCOMES:
Target Lesion Failure | 1 and 6 months
Bleeding rate according to BARC definition | 1, 6 and 12 months
Clinically driven target vessel revascularization | 1, 6 and 12 months
MACCE | 1, 6 and 12 months
  Cardiac death, stroke, myocardial infarction (Q wave and non Q wave) and TVR by non planned angioplasty or bypass graft
All deaths | 1, 6 and 12 months
Myocardial Infarction (MI) (Q wave and non Q wave) | 1, 6 and 12 months
Definite incidence of stent thrombosis | 1, 6 and 12 months
Clinically driven target lesion revascularization | 1, 6 and 12 months
Target lesion failure for patients >/= 80 years | 1, 6 and 12 months
Bleeding rate according to BARC definition for patients >/= 80 years | 1, 6 and 12 months
Target lesion failure for kidney failure patients (clearance < 30 ml/ min) | 1, 6 and 12 months
Bleeding Rate according to BARC definition for kidney failure patients (clearance < 30 ml/ min) | 1, 6 and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Jérôme Roncalli, Prof, Principal Investigator — CHU Toulouse, Hôpital Rangueil, TSA 50032, 31059 TOULOUSE Cedex 9
Locations (1):
- Chu Toulouse, Toulouse, France

REFERENCES:
- [Derived] Roncalli J, Godin M, Boughalem K, Shayne J, Piot C, Huret B, Belle L, Cayla G, Faurie B, Amor M, Karsenty B, Leclercq F. Paclitaxel Drug-Coated Balloon After Bare-Metal Stent Implantation, an Alternative Treatment to Drug-Eluting Stent in High Bleeding Risk Patients (The Panelux Trial). J Invasive Cardiol. 2019 Apr;31(4):94-100. doi: 10.25270/jic/18.00272. PMID 30927531